CLINICAL TRIAL: NCT04184999
Title: Evaluation of Intraoperative Use of Dexycu on the Signs and Symptoms of Dry Eye
Brief Title: Effect of Intraoperative Dexamethasone on Post-op Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SR Cornea Consultants (Other)
Responsible Party: Principal Investigator, Sanjay N Rao, MD, Principal Investigator, SR Cornea Consultants
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SRCC10
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Results first posted 2021-01-29 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Intervention Model Description: Randomized, controlled prospective study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intracameral dexamethasone 9% + postoperative topical prednisolone acetate (Experimental): dexamethasone intraocular suspension, 9% injected intracamerally at the time of cataract surgery + topical ophthalmic prednisolone acetate for 3 weeks post-operatively
  Interventions: Drug: dexamethasone intraocular suspension, 9%; Drug: Prednisolone Acetate 1% Oph Susp
- postoperative topical prednisolone acetate (Active Comparator): topical ophthalmic prednisolone acetate for 3 weeks post-operatively
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp

INTERVENTIONS:
Drug: dexamethasone intraocular suspension, 9% — single dose intracameral corticosteroid
  Other Names: Dexycu
  Arms: Intracameral dexamethasone 9% + postoperative topical prednisolone acetate
Drug: Prednisolone Acetate 1% Oph Susp — topical ophthalmic steroid drop

SUMMARY:
To compare the signs and symptoms of dry eye after cataract surgery between subjects randomized to receive intraoperative dexamethasone in addition to the use of a standard topical post-op treatment regimen.

DETAILED DESCRIPTION:
Forty patients requiring cataract surgery will be randomized to treatment of post-operative inflammation with a single intraoperative dexamethasone injection plus a standard course of topical ophthalmic corticosteroid drops or the standard treatment alone. Dry eye testing will be administered at baseline, 1 week and 3 weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing bilateral cataract surgery

Exclusion Criteria:

* central corneal staining with fluorescein and/or a tear film osmolarity of greater than 340 in either eye

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Rao, MD, Principal Investigator — SR Cornea Conslutants
Locations (1):
- Hauser Ross Surgical Center, Sycamore, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients scheduled to undergo bilateral cataract surgery 40 participants were enrolled, each eye was randomized to 2 different treatment groups (intracameral dexamethasone + postoperative topical prednisolone or postoperative topical prednisolone alone)
Pre-assignment Details: patients scheduled to undergo bilateral cataract surgery were randomly assigned to receive an intracameral injection of dexamethasone + a standard postoperative topical steroid regimen in one eye, and a standard postoperative topical steroid regimen in the other eye. Preoperative and postoperative signs of dry eye were compared between the two groups
Units Other Than Participants: eyes
Groups:
- Intracameral Dexamethasone + Postoperative Topical Prednisolone: dexamethasone intraocular suspension, 9% + topical ophthalmic prednisolone
  dexamethasone intraocular suspension, 9%: single dose intracameral corticosteroid
  Prednisolone Acetate: topical ophthalmic drop for 3 weeks
- Postoperative Topical Prednisolone: postoperative topical prednisolone for 3 weeks
Period: Overall Study
Arm/Group | Intracameral Dexamethasone + Postoperative Topical Prednisolone | Postoperative Topical Prednisolone
Started | 40; 40 eyes | 40; 40 eyes
3 Week Tear Film Osmolarity Testing | 40; 40 eyes | 40; 40 eyes
Completed | 40; 40 eyes | 40; 40 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: 40 participants undergoing bilateral cataract surgery were enrolled; 40 eyes were in the intracameral dexamethasone group and 40 eyes were in the standard postoperative regimen group
Units Other Than Participants: eyes
Groups:
- Intracameral Dexamethasone + Post-operative Topical Prednisolone: dexamethasone intraocular suspension, 9% + topical ophthalmic prednisolone
  dexamethasone intraocular suspension, 9%: single dose intracameral corticosteroid
  Prednisolone Acetate: topical ophthalmic drop
- Post-operative Topical Prednisolone: topical ophthalmic prednisolone acetate
  Prednisolone Acetate: topical ophthalmic drop
- Total: Total of all reporting groups
Arm/Group | Intracameral Dexamethasone + Post-operative Topical Prednisolone | Post-operative Topical Prednisolone | Total
Number analyzed (Participants) | 40 | 40 | 40
Number analyzed (eyes) | 40 | 40 | 80
Age, Categorical [Count of Units; unit: eyes] — 40 participants were enrolled, undergoing bilateral cataract surgery 40 eyes were in the intracameral dexamethasone group 40 eyes were in the standard postoperative regimen group
  eyes
    <=18 years | 1 | 1 | 2
    Between 18 and 65 years | 15 | 15 | 30
    >=65 years | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.49 (10.42) | 67.49 (10.42) | 67.49 (10.42)
Sex: Female, Male [Count of Units; unit: eyes]
  Female | 22 | 22 | 44
  Male | 18 | 18 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: eyes] — 40 participants were enrolled, each eye of each participant received was assigned to a different treatment group
  eyes
    United States | 40 | 40 | 80
Preoperative Tear Film Osmolarity [Mean (Full Range); unit: mOsmo/L] | 307.475 [292 to 320] | 307.775 [292 to 322] | 307.625 [292 to 322]

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Intraoperative Use of Dexycu on Tear Film Osmolarity at 3 Weeks Postoperatively
Description: Tear Film Osmolarity as measured on Tear Lab system; validated measure of Tear Film Osmolarity Osmolarity was reported in milliosmoles per liter (mOsmol/L)
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: mOsmol/L
Units Other Than Participants: eyes
Groups:
- Intracameral Dexamethasone: intracameral dexamethasone + postoperative prednisolone acetate for 3 weeks
- Postoperative Prednisolone Acetate: postoperative prednisolone acetate for 3 weeks
Arm/Group | Intracameral Dexamethasone | Postoperative Prednisolone Acetate
Number analyzed (Participants) | 40 | 40
Number analyzed (eyes) | 40 | 40
mOsmol/L | 311.15 [284 to 333] | 316.3 [286 to 335]
Statistical Analysis 1: Comparison: Intracameral Dexamethasone; Test type: Superiority; p < .01, ANOVA; F-Statistic = 207.4

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Intracameral Dexamethasone + Postoperative Prednisolone Acetate: intracameral dexamethasone 9% injection at the time of cataract surgery + standard postoperative prednisolone acetate regimen
- Postoperative Prednisolone Acetate Regimen: standard postoperative prednisolone acetate regimen
Arm/Group | Intracameral Dexamethasone + Postoperative Prednisolone Acetate | Postoperative Prednisolone Acetate Regimen
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT04184999/Prot_SAP_002.pdf
  • Informed Consent Form (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT04184999/ICF_000.pdf